CLINICAL TRIAL: NCT01404390
Title: An Open Label, Single Centre, Phase I Study of PI3K Inhibitor BAY80-6946 to Evaluate the Safety, Tolerability and Pharmacokinetics in Japanese Patients With Advanced or Refractory Solid Tumours
Brief Title: Japanese BAY80-6946 Monotherapy Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15205
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Neoplasms
Keywords: Phase I; Japanese
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY80-6946
- Arm 2 (Experimental)
  Interventions: Drug: BAY80-6946

INTERVENTIONS:
Drug: BAY80-6946 — 0.4mg/ kg, iv, day 1,8 and 15, every 28 days
  Arms: Arm 1
Drug: BAY80-6946 — 0.8mg/ kg, iv, day 1,8 and 15, every 28 days
  Arms: Arm 2

SUMMARY:
This study will be conducted as an open label, single centre, Phase I study of PI3K (phosphatidyl inositol 3 kinase) inhibitor BAY80-6946 in Japanese patients with advanced or refractory solid tumours. The eligible subjects will be dosed intravenously at Day 1, Day 8 and Day 15 with three weeks on and one week off in each treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Japanese patients, who are at least 20 years of age
* Histological or cytological documentation of non-hematologic, malignant solid tumours, excluding primary brain or spinal tumours, with no past or current involvement in the central nervous system (CNS)
* At least one measurable lesion or evaluable disease according to RECIST (version 1.1)
* Eastern Cooperative Oncology performance status (ECOG-PS) of 0 or 1
* Life expectancy of at least 12 weeks
* Advanced or refractory solid tumours not amenable to standard therapy, at the first screening examination/visit

Exclusion Criteria:

* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of first study treatment. Patients must have recovered from the toxic effects of the previous anti-cancer chemotherapy or immunotherapy by the investigator (with the exception of alopecia).
* Radiotherapy to target lesions during study or within 4 weeks of first study treatment
* Investigational drug therapy outside of this trial during or within 4 weeks of first study treatment
* Current diagnosis of Type I or II diabetes mellitus or fasting blood glucose level >125 mg/dL at screening, and/or HbA1c>/= 6.5%
* Past and current histories of cardiac disease congestive heart failure > New York Heart Association (NYHA) Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset of angina within 3 months prior to study entry or unstable angina or ventricular cardiac arrhythmias requiring anti-arrhythmic therapy
* Active and clinically serious infections >Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 4.03)
* Uncontrolled hypertension defined as systolic blood pressure >150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* Patients undergoing renal dialysis
* Pregnant or breast feeding women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08-18 (Actual); Primary Completion 2012-03-22 (Actual); Study Completion 2012-07-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 169 days
Maximum drug concentration in plasma after single dose administration (Cmax) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15, 0 - 8 hours in Cycle3 Day15
Cmax divided by dose (mg) per kg body weight (Cmax,norm) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15, 0 - 8 hours in Cycle3 Day15
Cmax divided by dose (mg) (Cmax/D) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15, 0 - 8 hours in Cycle3 Day15
Area under the concentration-time curve time 0 to 8 hours (AUC(0-8)) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15, 0 - 8 hours in Cycle3 Day15
Area under the concentration-time curve from time 0 to 25 hours (AUC(0-25)) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15
AUC(0-25) divided by dose (mg) per kg body weight (AUC(0-25)norm) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15
AUC(0-25) divided by dose (mg) (AUC(0-25)/D) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15
AUC from time 0 to last data point (AUC(0-tlast)) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15
Time to maximum drug concentration in plasma (tmax) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15, 0 - 8 hours in Cycle3 Day 15

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve of (AUC) of BAY80-6946 | 0 - 168 hours in Cycle1 Day1
Half-life associated with terminal slope of drug in plasma (t1/2) | 0 - 168 hours in Cycle1 Day1
Mean residence time of drug in plasma (MRT) | 0 - 168 hours in Cycle1 Day1
Total body clearance of drug from plasma (CL) | 0 - 168 hours in Cycle1 Day1
Volume of drug distribution during terminal phase after single dose administration (Vz) | 0 - 168 hours in Cycle1 Day1
Volume of drug distribution during steady state after single dose administration (Vss) | 0 - 168 hours in Cycle1 Day1
Accumulation ratio calculated from AUC(0-8) after multiple dosing and AUC(0-8) after single dosing (RAAUC(0-8)) | 0 - 8 hours in Cycle3 Day15
Accumulation ratio calculated from AUC(0-25) after multiple dosing and AUC(0-25) after single dosing (RAAUC(0-25)) | 0 - 25 hours in Cycle1 Day15
Accumulation ration calculated from Cmax after multiple dosing and Cmax after single dosing (RACmax) | 0 - 168 hours in Cycle1 Day1, 0 - 25 hours in Cycle1 Day15
Overall tumor response rate | 176 days
  Proportion of subjects with confirmed complete and partial response
Overall disease control rate | 176 days
  Proportion of subjects who had a best response rating of complete response, partial response or stable disease
Time to progression of cancer growth | 176 days
Progression-free survival time | 176 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Kashiwa, Chiba, Japan

REFERENCES:
- [Derived] Doi T, Fuse N, Yoshino T, Kojima T, Bando H, Miyamoto H, Kaneko M, Osada M, Ohtsu A. A Phase I study of intravenous PI3K inhibitor copanlisib in Japanese patients with advanced or refractory solid tumors. Cancer Chemother Pharmacol. 2017 Jan;79(1):89-98. doi: 10.1007/s00280-016-3198-0. Epub 2016 Dec 3. PMID 27915408